CLINICAL TRIAL: NCT02760667
Title: A Phase II Study of Induction Chemotherapy Followed by Surgical Treatment in Locally Advanced Oropharyngeal And Supraglotic Cell Carcinoma
Brief Title: Induction Chemotherapy Followed by Surgery for Locally Advanced Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Robert Siegel, Professor of Medicine, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWU-MFA Head and Neck Protocol
Record Dates: First submitted 2016-04-08; First posted 2016-05-04 (Estimated); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer
Keywords: Oropharyngeal cancer; Laryngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms | interventions — Cisplatin; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Induction Therapy with 3 cycles (Experimental): Cisplatin 75mg/m2 IV and Taxotere 75mg/m2 every 3 weeks for 3 cycles (Induction Chemotherapy) followed by surgical treatment
  Interventions: Drug: Cisplatinum; Drug: Docetaxel; Drug: Carboplatin; Procedure: Transoral Robotic Assisted Surgery

INTERVENTIONS:
Drug: Cisplatinum — Cisplatin 75mg/m2 every 3 weeks for a maximum of 3 cycles during the induction phase
  Other Names: Cisplatin
Drug: Docetaxel — Docetaxel 75mg/m2 every 3 weeks for a maximum of 3 cycles during the induction phase
  Other Names: Taxotere
Drug: Carboplatin — Carboplatin AUC=5 every 3 weeks for a maximum of 3 cycles during the induction phase (if subject are unable to tolerate cisplatin)
  Other Names: Paraplatin
Procedure: Transoral Robotic Assisted Surgery — TORS will be performed for the patients who responded to the induction treatment (80% reduction)
  Other Names: TORS

SUMMARY:
The objective of this study is to assess the efficacy of induction chemotherapy followed by transoral surgical treatment and neck dissection, in definitive management of moderately advanced oropharyngeal squamous cell carcinoma. The surgical treatment will carry out Transoral Robotic Surgery (TORS) or Transoral Laser Microsurgery (TLM) for the primary tumor, and neck dissection for the management of cervical lymph nodes.

The primary outcome measure will be disease specific survival (DSS). The secondary oncologic outcome measures will be locoregional control, relapse free survival, overall survival, and Quality of Life (QOL).

DETAILED DESCRIPTION:
The current standard of care for advanced (stage III and IV) oropharyngeal squamous cell carcinoma are concomitant chemoradiation, or surgery followed by adjuvant radiation therapy with or without concomitant chemotherapy. These approaches have persistent and significant lifelong side effects and sequella related to treatment, and in particular radiotherapy. The side effects of radiotherapy (augmented with concomitant chemotherapy) include soft tissue fibrosis, loss of salivary function, dry mouth, life long disturbed taste function, poor dental health with rapidly decaying teeth, dysfunction of swallowing, significant loss of the mobility of the base of tongue and pharyngeal constrictors, loss of laryngeal elevation, esophageal stricture, and at times severe side effects such as soft tissue necrosis or osteoradionecrosis of the mandible. About 10% of the patients undergoing chemoradiation for oropharyngeal cancer develop long term swallowing dysfunction with feeding tube dependency. As a result , patient's quality of life (QOL) is adversely affected. Improvements in the side effect profile of treatment, the functional outcome, and the QOL remain very important areas of advancement in treating this patient population. Improvements in functional outcome need to be achieved while maintaining or improving the oncologic outcome and cure rates for cancer, compared to the standard of care.

Use of new Taxane based chemotherapy along with Platinum drugs (Cisplatin and Carboplatin) in high dose neoadjuvant setting, coupled with novel minimally invasive Transoral Laser Microsurgery (TLM) and Transoral Robotic Assisted Surgery (TORS), allows potential for improved oncologic outcome as well as avoidance of long term sequalla of high dose radiation therapy to head and neck. These transoral surgical approaches (TLM and TORS) provide improved functional outcome compared with traditional open composite resections and complex reconstructive algorithms for oropharynx. TLM and TORS are currently in clinical use for early (stage T1 and T2 with N0 or N+ve) oropharyngeal cancer.

An area not adequately or at all investigated in treating moderately advanced oropharyngeal cancer is combining neoadjuvant high dose chemo-induction followed by minimally invasive transoral surgery (TLM and TORS) and neck dissection as the definitive treatment.

This approach has the potential for far improved functional outcome by avoiding short and more importantly long term and permanent sequella of radiation therapy in oropharyngeal cancer treatment. This approach is a new paradigm in treatment of oropharyngeal cancer, and can significantly improve the functional outcome of cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven squamous cell carcinoma of the oropharynx (tonsil, base of tongue, vallecula, soft palate) and supraglottis.
* Stages III (T1N1, T2N1, T3N0, T3N1) and stage IVA (T1N2, T2N2, T3N2, very select earlyT4) disease not previously treated with any method (Surgery, Radiation or Chemotherapy)
* No evidence of distant metastatic disease
* Fit for surgery and primary tumor assessed surgically resectable (by surgical PI) via transoral approach
* Age > 18 years
* Karnofsky performance status > 60%, or ECOG < 2
* ANC > 2,000, platelets > 100,000 and calculated creatinine clearance >50 cc/min
* Signed study specific consent form
* Protocol begins within 4 weeks of biopsy and within 3 weeks of the latest medical imaging.

  * No other malignancies except cutaneous basal or squamous cell cancer within the last 5 years
  * Patients must have measurable disease based on RECIST.
* Men and women of child bearing potential must agree to use effective contraception while on the study, and women must have a negative pregnancy test, and not be lactating.

Exclusion Criteria:

* Patients with advanced T4 cancer judged unresectable by transoral approach by surgical PI.
* Patients with N3 disease (Stage IVB).
* Patients with distant metastatic disease (Stage IVC).
* Patients with radiologically positive neck nodes with radiological evidence of extracapsular nodal tumor invasion.
* Patients having anatomy not allowing transoral access and exposure for surgery(Judged by the surgical PI at the time of biopsy under general anesthesia)
* Patients with prior head and neck cancer at any time (other than basal or squamous cell cancer of the skin)
* Coexistent second malignancy or history within 5 years of prior malignancy (other than basal or squamous cell cancer of the skin or curatively treated Stage I carcinoma of the cervix) renders the patient ineligible.
* Patients with peripheral neuropathy >/= grade 1 will not be eligible for the study.
* Patients who have had prior Taxanes or Cisplatin
* Patients with concurrent infection are not eligible. All patients must be afebrile for at least 3 days prior to start of therapy unless fever is due to tumor.
* Patients with coexisting medical illness of a severity that might interfere with treatment or follow-up, or who do not have the ability to give informed consent.
* Patients who have received prior radiation therapy, surgery and chemotherapy for the tumor being treated.
* Patients must not be receiving any other investigational agent while on the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease specific survival (DSS) | 3 years
  this parameter is a number will tell the chances of staying free of the head and neck cancer after the study treatment.

SECONDARY OUTCOMES:
Relapse-free survival | 3 years
  Considering the length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer.
Overall survival | 3 years
  Measure of the length of time from either the date of diagnosis or the start of treatment for a disease that patients diagnosed with the disease are still alive.
EORTC QLQ-C30 | 3 years
  EORTC QLQ C-30 questionnaire will be administered at baseline (prior to induction chemotherapy), at the end of the 3rd cycle of induction treatment , after surgery, 3 months post-surgery for 1 year and every 6 months thereafter (years 2 and 3)
EORTC QLQ-H&N35 | 3 years
  EORTC QLQ H&N35 questionnaire will be administered at baseline (prior to induction chemotherapy), at the end of the 3rd cycle of induction treatment , after surgery, 3 months post-surgery for 1 year and every 6 months thereafter (years 2 and 3)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Siegel, M.D., Study Chair — George Washington University
Locations (1):
- George Washington University-Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No